CLINICAL TRIAL: NCT01167257
Title: Comparative Study of the Efficacy and Safety of Liposome Encapsulated Botulinum Toxin-A (Lipotoxin) Versus Normal Saline Instillation in Treatment of Patients With Refractory Overactive Bladder Syndrome
Brief Title: Effects and Safety of Liposome Encapsulated Botulinum Toxin A for Overactive Bladder Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Department of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCGHUROL001
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Detrusor overactivity; Liposome; Botulinum toxin A
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental arm (Experimental): Liposome encapsulated BoNT-A ( mixed BOTOX 200 U/10 mL in Liposome 80 mg/40 mL) in single intravesical instillation
  Liposome encapsulated botulinum toxin A'
  Interventions: Drug: Liposome encapsulated botulinum toxin A
- Control arm (Placebo Comparator): Normal saline 50 mL in single intravesical instillation
  Normal saline instillation'
  Interventions: Drug: Normal saline instillation

INTERVENTIONS:
Drug: Liposome encapsulated botulinum toxin A — Liposome encapsulated BoNT-A ( mixed BOTOX 200 U/10 mL water in Liposome 80 mg/40 mL water) in single intravesical instillation, one time treatment at the treatment day
  Other Names: Lipotoxin
  Arms: Experimental arm
Drug: Normal saline instillation — Normal saline (BoNT-A/NS) 50 mL in single intravesical instillation
  Other Names: N/S
  Arms: Control arm

SUMMARY:
Overactive bladder (OAB) is a bothered symptom syndrome. Traditional medication for OAB is antimuscarinic agent. However, adverse events such as dry mouth, constipation, blurred vision, and dizziness may prohibit patient to take this drug for OAB. Intravesical botulinum toxin A (BoNT-A) is a novel treatment however, BoNT-A can cause acute urinary retention and large postvoid residual. In this grant we will evaluate liquid liposome delivery of BoNT-A (Liposome encapsulated BoNT-A) into the bladder without the need for cystoscopic-guided needle injection for refractory OAB.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a symptom syndrome characterized by urgency frequency with or without urgency incontinence, usually no metabolic or anatomical disorders can be found and it may have great impact on quality of life. Traditional medication for OAB is antimuscarinic agent which targets at the muscarinic receptors. There are several adverse events such as dry mouth, constipation, blurred vision, and dizziness related to antimuscarinics, therefore, some patients cannot tolerated this treatment. Intravesical botulinum toxin A (BoNT-A) has recently emerged as novel treatment for OAB refractory to antimuscarinics, however, BoNT-A injection can cause acute urinary retention and large postvoid residual. Urinary tract infection usually occurred following large postvoid residual and urinary retention. If we can deliver BoNT-A through the urothelium to the suburothelial space, but not into the detrusor layer, we might have therapeutic effects on the urothelial sensory nerves without compromising the detrusor contractility. This treatment will enable us to prevent the undesired detrusor underactivity after BoNT-A injection, especially in the elderly patients who had impaired detrusor contractility and OAB. Liposomes are vesicles, composed of concentric phospholipid bilayers separated by aqueous compartments. Because liposomes adsorb to cell surfaces and fuse with cells, they are being used as vehicles for drug delivery and gene therapy. In this grant we will evaluate liquid liposome delivery of BoNT-A (Liposome encapsulated BoNT-A) into the bladder without the need for cystoscopic-guided needle injection for refractory OAB, and study the mechanism of action of intravesical liposomal drug delivery. If successful, we will leverage our technology transfer expertise and bring the science from the bench top to the bed side to apply for a physician sponsored Investigational New Drug (IND) trial using liposome-BoNT in patients with OAB or DO.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with age of 20 years old or above
2. Patients with symptoms of urgency frequency and/or urge incontinence and a urgency severity scale (USS) of at least 2, with or without urodynamically proven detrusor overactivity (DO) (defined by the International Continence Society (ICS) recommendation as: spontaneous detrusor contraction occurring during bladder filling phase or occurring before uninhibited detrusor contraction voiding at bladder capacity in the urodynamic study)
3. Free of active urinary tract infection
4. Free of bladder outlet obstruction on enrollment
5. Free of overt neurogenic bladder dysfunction
6. Having been treated with antimuscarinic agents for at least 4 weeks without effect or with intolerable adverse effects
7. Patient has not been treated with bladder surgery for OAB, such as enterocystoplasty, that might affect the therapeutic effect of test drug
8. Patient can record voiding diary for the urinary frequency and urgency
9. Patient or his/her legally acceptable representative has signed the written informed consent form

Exclusion Criteria:

1. Use of antimuscarinic agent and effective in treatment of lower urinary tract symptoms
2. Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up
3. Patients with bladder outlet obstruction on enrollment
4. Patients with postvoid residual >150 mL
5. Patients with uncontrolled confirmed diagnosis of acute urinary tract infection
6. Patients have laboratory abnormalities at screening including:

   Alanine aminotransferase (ALT) >3 x upper limit of normal range Aspartate aminotransferase (AST) >3 x upper limit of normal range Patients have abnormal serum creatinine level >2 x upper limit of normal range
7. Patients with any contraindication to be urethral catheterization during treatment
8. Female patients who is pregnant, lactating, or with child-bearing potential without contraception.
9. Myasthenia gravis, Eaton Lambert syndrome.
10. Patients with any other serious disease considered by the investigator not suitable for general anesthesia or in the condition to enter the trial
11. Patients participated investigational drug trial within 1 month before entering this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital and Tzu Chi University; Yao-Chi Chuang, M.D., Principal Investigator — Department of Urology, Chang Gung Memorial Hospital, Kaohsiung, Taiwan
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10 mL in Liposome 80 mg/40 mL) in single intravesical instillation
  Liposome encapsulated botulinum toxin A: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10 mL water in Liposome 80 mg/40 mL water) in single intravesical instillation, one time treatment at the treatment day
- Control Arm: Normal saline 50ml in single intravesical instillation
  Normal saline instillation: Normal saline (BoNT-A/NS) 50ml in single intravesical instillation
Period: Overall Study
Arm/Group | Experimental Arm | Control Arm
Started | 31 | 31
Completed | 28 | 28
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrew consent | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental Arm: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10 mL in Liposome 80mg/40ml) in single intravesical instillation
  Liposome encapsulated botulinum toxin A: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10 mL water in Liposome 80 mg/40 mL water) in single intravesical instillation, one time treatment at the treatment day
- Control Arm: Normal saline 50 mL in single intravesical instillation
  Normal saline instillation: Normal saline (BoNT-A/NS) 50ml in single intravesical instillation
- Total: Total of all reporting groups
Arm/Group | Experimental Arm | Control Arm | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.43 (12.49) [48 to 82] | 65.81 (14.48) [38 to 73] | 65.12 (13.49) [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 15 | 33
  Male | 13 | 16 | 29
Region of Enrollment [Number; unit: participants]
  Taiwan | 31 | 31 | 62
Associated medical conditions [Number; unit: participants]
  Diabetes Mellitus | 3 | 9 | 12
  Hypertension | 5 | 12 | 17
  Pelvic surgery | 0 | 1 | 1
  Other disease | 1 | 1 | 2
  Non disease | 22 | 8 | 30
Background or Prior disease [Number; unit: participants]
  Any prior disease | 31 | 31 | 62
  None | 0 | 0 | 0
Prior therapy [Number; unit: participants]
  Prior therapy taken | 29 | 29 | 58
  None | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of the Total Frequency Per 3 Days
Description: Efficacy:
  Mean change of the total frequency per 3 days from baseline to 4 weeks after the treatment day based on the 3-day voiding diary.
  Change = Week 4 minus Baseline value
Time Frame: Baseline to 4 weeks after initial treatment
Population: Control arm: subject number S025 was removed from analysis for not meeting the requirement for analysis, thus control arm 27 subjects
Measure: Mean (95% Confidence Interval); unit: Frequency per 3 days
Groups:
- Control Arm: Normal saline 50 mL in single intravesical instillation
  Normal saline instillation: Normal saline (BoNT-A/NS) 50 mL in single intravesical instillation
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 28 | 27
Frequency per 3 days | -4.64 [-7.46 to -1.82] | -0.19 [-2.98 to 2.61]

2. Secondary Outcome: Mean Change of the Urgency Episodes Per 3 Days
Description: Efficacy:
  Mean change of the Urgency episodes per 3 days from baseline to 4 weeks after the treatment day based on the 3-day voiding diary.
  Change = Week 4 minus Baseline value
Time Frame: Baseline to 4 weeks after initial treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Frequency per 3 days
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 28 | 27
Frequency per 3 days | -7.43 [-11.68 to -3.18] | -3.43 [-7.30 to 0.45]

3. Secondary Outcome: Mean Change of the Urgency Urinary Incontinence (UUI) Per 3 Days
Description: Efficacy:
  Mean change of the urgency urinary incontinence (UUI) per 3 days from baseline to 4 weeks after the treatment day based on the 3-day voiding diary.
  Change = Week 4 minus Baseline value
Time Frame: Baseline to 4 weeks after initial treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Frequency per 3 days
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 28 | 27
Frequency per 3 days | 0.43 [-3.33 to 4.19] | 0.56 [-1.27 to 2.38]

4. Secondary Outcome: Net Change of the Overactive Bladder Symptom Score (OABSS)
Description: Efficacy:(measured the net change of variables from baseline to 1 month) Overactive bladder symptom score (OABSS) The OABSS is a 4-item questionnaire developed to evaluate OAB symptoms. The maximal scores are 2, 3, 5 and 5 for daytime frequency, nighttime frequency, urgency and urgency in continence, respectively.
  The OABSS range = 0 to 15 ((asymptomatic to very symptomatic). Change = Week 4 minus Baseline value
Time Frame: Baseline to 4 weeks after initial treatment
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Experimental Arm: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10ml in Liposome 80 mg/40 mL) in single intravesical instillation
  Liposome encapsulated botulinum toxin A: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10 mL water in Liposome 80 mg/40 mL water) in single intravesical instillation, one time treatment at the treatment day
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 28 | 28
units on a scale | -1.86 [-2.96 to -0.76] | -0.75 [-2.01 to 0.51]

5. Secondary Outcome: Net Change of the Functional Bladder Capacity (FBC)
Description: Efficacy:(measured the net change of variables from baseline and 1 month) Functional bladder capacity (FBC) Change = Week 4 minus Baseline value
Time Frame: Baseline to 4 weeks after initial treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 28 | 27
mL | -12.86 [-45.79 to 20.08] | 18.15 [-16.37 to 52.67]

6. Secondary Outcome: Net Change of the Maximum Flow Rate (Qmax)
Description: Efficacy:(measured the net change of variables from baseline and 1 month) Maximum flow rate (Qmax) Change = Week 4 minus Baseline value
Time Frame: Baseline to 4 weeks after initial treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mL/s
Groups:
- Experimental Arm: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10 mL in Liposome 80 mg/40 mL) in single intravesical instillation
  Liposome encapsulated botulinum toxin A: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10 mL water in Liposome 80 mg/40 Ll water) in single intravesical instillation, one time treatment at the treatment day
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 28 | 27
mL/s | 0.11 [-2.02 to 2.25] | -0.84 [-4.30 to 2.62]

7. Secondary Outcome: Net Change of the Postvoid Residual Volume (PVR)
Description: Efficacy:(measured the net change of variables from baseline and 1 month) Postvoid residual volume (PVR) Change = Week 4 minus Baseline value
Time Frame: Baseline and 1 month after initial treatment
Measure: Median (Inter-Quartile Range); unit: mL
Groups:
- Experimental Arm: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10 mL in Liposome 80 mg/40 mL) in single intravesical instillation
  Liposome encapsulated botulinum toxin A: Liposome encapsulated BoNT-A ( mixed BOTOX 200 U/10 mL water in Liposome 80 mg/40 mL water) in single intravesical instillation, one time treatment at the treatment day
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 28 | 28
mL | -2.65 [-20.13 to 14.84] | -2.31 [-19.43 to 14.81]

8. Secondary Outcome: Net Change of the Urgency Severity Score (USS) Within 3 Days
Description: Efficacy:(measured the net change of variables from baseline and 1 month) Urgency severity score (USS) within 3 days. The USS have 1-point scale ranging from 0 to 4. The USS grades urgency per toilet void as none, mild, moderate or severe.
Time Frame: Baseline to 4 weeks after initial treatment
Measure: Number; unit: participants
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 28 | 28
participants
  Improved | 11 | 4
  No change | 16 | 20
  Worsen | 1 | 4

9. Secondary Outcome: Net Change of the Global Response Assessment (GRA)
Description: Efficacy:(measured the net change of variables from baseline and 1 month) The Global response assessment (GRA) have seven point scale is centered at zero (no change): markedly worse; moderately worse; slightly worse; no change; slightly improved; moderately improved; and markedly improved.
Time Frame: Baseline to 4 weeks after initial treatment
Measure: Number; unit: participants
Arm/Group | Experimental Arm | Control Arm
Number analyzed (Participants) | 28 | 28
participants
  Improved | 21 | 19
  No change | 7 | 9

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Experimental Arm: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10 mL in Liposome 80 mg/40 mL) in single intravesical instillation
  Liposome encapsulated botulinum toxin A'
  Liposome encapsulated botulinum toxin A: Liposome encapsulated BoNT-A (mixed BOTOX 200 U/10 mL water in Liposome 80 mg/40 mL water) in single intravesical instillation, one time treatment at the treatment day
- Control Arm: Normal saline 50 mL in single intravesical instillation
  Normal saline instillation'
  Normal saline instillation: Normal saline (BoNT-A/NS) 50 mL in single intravesical instillation
Arm/Group | Experimental Arm | Control Arm
Serious Adverse Events (participants affected / at risk) | 1/31 | 2/31
Other Adverse Events (participants affected / at risk) | 10/31 | 16/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm (N=31) | Control Arm (N=31)
Hyponatremia (General disorders) | 0 | 1
Right Knee osteoarthritis (General disorders) | 1 | 0
C-spine whiplash injury with radiculopathy (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm (N=31) | Control Arm (N=31)
Cervical spondylosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foreign body in conjunctival SAC (Eye disorders) | 1 | 0
Diabetes mellitus (Endocrine disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Unspecified otitis media (Ear and labyrinth disorders) | 1 | 0
Chronic mastoiditis (Reproductive system and breast disorders) | 1 | 0
Dizziness and giddiness (General disorders) | 1 | 0
Abdominal fullness pain (Gastrointestinal disorders) | 1 | 0
Respiratory infection upper tract (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Couch (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Unspecified local infections of skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 0 | 1
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fracture of ankle (Musculoskeletal and connective tissue disorders) | 0 | 1
Traumatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture of clavicle (Musculoskeletal and connective tissue disorders) | 0 | 1
Paralysis (Nervous system disorders) | 0 | 1
Contusion (Skin and subcutaneous tissue disorders) | 0 | 1 — Contusion of face, scalp, neck except eye
Functional disorder of stomach disturbance irritation (Gastrointestinal disorders) | 0 | 1
Herpes zoster (Skin and subcutaneous tissue disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Oral ulcer (General disorders) | 0 | 1
Blepharitis (Eye disorders) | 0 | 1
Rhinitis (General disorders) | 0 | 2
Dermatophytosis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes